CLINICAL TRIAL: NCT00365196
Title: Hostility Reduction and Autonomic Control of the Heart
Brief Title: Hostility Reduction Program to Improve Autonomic Regulation of the Heart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Richard P. Sloan, Columbia University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 399; R01HL063872-04 (NIH)
Record Dates: First submitted 2006-08-16; First posted 2006-08-17 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2007-12

CONDITIONS: Hostility; Coronary Arteriosclerosis
Keywords: Autonomic Nervous System
MeSH Terms: conditions — Coronary Artery Disease

INTERVENTIONS:
Behavioral: CBT Hostility Reduction Program

SUMMARY:
Individuals who experience high hostility levels may be more prone to developing coronary artery disease (CAD) than individuals who experience low hostility levels. This study will evaluate the effectiveness of a hostility reduction treatment program on the body's ability to regulate heart activity in individuals with high levels of hostility.

DETAILED DESCRIPTION:
CAD is caused by a narrowing of the blood vessels that supply blood and oxygen to the heart. It is the leading cause of death in the United States. Recent evidence has suggested that individuals with increased hostility levels have a higher risk of developing CAD than individuals with lower hostility levels. The autonomic nervous system (ANS), the involuntary part of the nervous system that is responsible for controlling the body's internal environment in a coordinated manner, may play a role in CAD development. High levels of hostility may elevate ANS activity and increase the release of certain hormones, which in turn may lead to hardening of the arteries and CAD. Cognitive behavioral therapy (CBT) has been effective for treating individuals with hostility. Through CBT, individuals develop coping skills to deal with their anger. This study will evaluate the effect of a CBT hostility reduction treatment program on ANS heart regulation and overall CAD risk in individuals with high levels of hostility.

This study will enroll individuals with high levels of hostility. At an initial screening visit, potential participants will partake in interviews and complete questionnaires to assess hostility levels. Eligible participants will then undergo 24-hour continuous electrocardiogram (ECG) monitoring and will complete questionnaires about their surroundings and any hostility experienced during the 24-hour period. They will also undergo psychophysiological testing, in which responses to a variety of stress-inducing situations will be monitored. Participants will then be randomly assigned to either a 12-week CBT hostility reduction treatment program or a 12-week wait list control group. Participants in the CBT program will attend weekly 75-minute therapy sessions, which will focus on relaxation, stress reduction, behavior management, and development of social, communication, and coping skills. Hostility levels will be documented each day in a diary. Participants in the wait list control group will not take part in any therapy sessions for the initial 12 weeks. At Week 12, baseline evaluations will be repeated for all participants. The waitlist control group will then begin the 12-week CBT program. All participants will attend a 6-month follow-up visit for repeat testing.

ELIGIBILITY:
Inclusion Criteria:

* In good general health
* Experiences a high level of hostility according to the Spielberger Trait Anger Scale and Cook Medley Scale (greater than 1 standard deviation for each scale)
* English speaking

Exclusion Criteria:

* Psychiatric disorder
* Currently taking psychiatric medications
* Currently taking cardioactive medications
* Medical condition that affects the ANS
* Currently taking medications that affect the cardiovascular system

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150
Dates: Start 1999-12; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Cardiac autonomic regulation (measured at Week 12 and at 6-month follow-up evaluation)

CONTACTS AND LOCATIONS:
Overall Officials: Richard P. Sloan, PhD, Principal Investigator — Columbia University

REFERENCES:
- [Derived] Sloan RP, Shapiro PA, DeMeersman RE, Bagiella E, Brondolo EN, McKinley PS, Crowley O, Zhao Y, Schwartz JE, Myers MM. Impact of aerobic training on cardiovascular reactivity to and recovery from challenge. Psychosom Med. 2011 Feb-Mar;73(2):134-41. doi: 10.1097/PSY.0b013e31820a1174. Epub 2011 Jan 21. PMID 21257979